CLINICAL TRIAL: NCT05586373
Title: Use of Ibuprofen Versus Dipyrone in Preeclampsia Submitted to C-section: Randomized Clinical Trial
Brief Title: Ibuprofen vs Dipyrone After C-section in Preeclampsia
Acronym: DIPROFEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, MD PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIPROFEN
Record Dates: First submitted 2022-10-10; First posted 2022-10-19 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; postpartum period; NSAIDs; acute kidney injury; cesarean section; analgesia
MeSH Terms: conditions — Pre-Eclampsia; Acute Kidney Injury; Agnosia | interventions — Ibuprofen; Dipyrone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Ibuprofen 400mg 6/6h, oral, maximum 5 days
  Interventions: Drug: medication 1
- Group 2 (Experimental): Dipyrone 1g 6/6h, oral, maximum 5 days
  Interventions: Drug: medication 2

INTERVENTIONS:
Drug: medication 1 — Ibuprofen pills, identical to the intervention (dipyrone pills), will be administered every 6 hour for a maximum of five days
  Other Names: Ibuprofen 400 mg
  Arms: Group 1
Drug: medication 2 — Dipyrone pills, identical to the intervention (ibuprofen pills), will be administered every 6 hour for a maximum of five days
  Other Names: Dipyrone 1g
  Arms: Group 2

SUMMARY:
The goal of this randomized, triple-masked clinical trial is to compare the effectiveness and safety of the use of ibuprofen versus dipyrone for postoperative analgesia in postpartum women with preeclampsia undergoing cesarean section.

The main question it aims to answer are:

* Postoperative pain is similar;
* The frequency of acute kidney injury is similar.

Researchers will compare one group that will receive dipyrone and the other group that will receive ibuprofen to see if Postoperative pain are different between groups or development of acute kidney injury each group is different.

DETAILED DESCRIPTION:
Specific objectives

In postpartum women with preeclampsia undergoing cesarean section randomized to receive treatment with ibuprofen versus dipyrone for postoperative analgesia, compare:

primary outcomes

1. Postoperative pain (mild, moderate, severe by visual analogue scale)
2. Development of acute kidney injury (serum creatinine 1.5 to 1.9 times baseline, or increase in serum creatinine by ≥0.3 mg/dL, or decrease in urine output to <0.5 mL/kg/ hour for six to 12 hours).

secondary outcomes

1. Average reduction of visual analogue scale scores;

2 Reduction of mean scores by algometer;

3. Need for rescue analgesic;

4. User satisfaction with the Likert scale;

5. Basic laboratory tests and their evolution: urea, creatine, uric acid, saline, potassium and chlorine, lactic dehydrogenase (DHL), aspartate transferase (AST), alanine transferase (ALT), total and fractions bilirubin and plaque;

6. Evolution of blood pressure in the puerperium;

7. Number of hypertensive peaks;

8. Need for maintenance antihypertensive treatment and number of drugs;

9. Allergic reactions;

10. Gastrointestinal side effects;

11. Time between postoperative and unassisted ambulation;

12. Length of hospital stay;

13. Compound maternal morbidity (eclampsia, acute weight edema, HELLP, difficulty hypertension, intracranial hemorrhage, renal function control and others);

14. Maternal death;

15. Costs related to analgesic medications.

The sample is 74 patients randomized into two groups: one group that will receive dipyrone and the other group that will receive ibuprofen. Randomization for the two groups will be performed according to a list of random numbers drawn up for that purpose by an employee who does not be involved with data collection, to ensure confidentiality in the allocation. From this list, sealed envelopes will be prepared, numbered sequentially, with each number, according to the randomization table, corresponding to the patient's group (dipyrone or ibuprofen).

For statistical analysis of the data, the domain statistical program will be used public Epi-info version 7, or higher versions. Tables will be distributed frequency distribution for categorical variables, calculating the mean and standard deviation of quantitative variables. Then, contingency tables will be used to determine the association of the independent variable (Ibuprofen versus dipyrone) with the dependent variables (Biological characteristics, obstetric features, Maternal clinical parameters at admission and during hospitalization, Maternal laboratory tests at the time of admission). For determination of the strength of association will be calculated as a measure of the risk (RR) and its 95% confidence interval. All p values will be two-tailed and in all stages of the analysis will be considered a level of significance 5%.

ELIGIBILITY:
Inclusion Criteria:

* Puerperal women from 14 years of age diagnosed with preeclampsia with signs of severity Immediate postoperative period;
* Delivery attended at the Maternity from Instituto de Medicina Integral Prof Fernando Figueira.

Exclusion Criteria:

* Acute kidney disease (serum creatinine 1.5 to 1.9 times baseline, or increase in serum creatinine by ≥0.3 mg/dL, or decrease in urine output to <0.5 mL/kg/hour for six to 12 hours)
* Chronic kidney disease;
* Diabetes mellitus;
* Collagenoses;
* Sickle cell anemia;
* Patients who presented bleeding in the pre, trans and immediate postpartum periods;
* Antepartum or puerperal sepsis;
* Known contraindications to the use of NSAIDs and dipyrone;

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | from 24 after delivery to 48 hours
  Postoperative pain (mild, moderate, severe by visual analogue scale)
Development of acute kidney injury | from 24 after delivery to 48 hours
  Development of acute kidney injury (serum creatinine 1.5 to 1.9 times baseline, or increase in serum creatinine by ≥0.3 mg/dL, or decrease in urine output to <0.5 mL/kg/ hour for six to 12 hours).

SECONDARY OUTCOMES:
Mean reduction of pain scores by visual analogue scale; | from 24 after delivery to 48 hours
  Mean reduction of pain scores by visual analogue scale;
Mean reduction in pain scores assessed by algometer | from 24 after delivery to 48 hours
  Mean reduction in pain scores assessed by algometer
need for rescue analgesic therapy; | from 24 after delivery to 48 hours
  Quantify the number of times analgesic medication was requested, in addition to what is being offered in the study
User satisfaction level | from 24 after delivery to 48 hours
  Likert scale, used in questionnaires, Participants choose from a variety of possible responses to a specific question or statement; responses usually include "strongly agree", "agree", "neutral", "disagree" and "strongly disagree".
urea dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, urea measured in mg/dl at admission and up to 48 hours after admission.
aspartate transferase dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, aspartate transferase dosage measured in mg/dl at admission and up to 48 hours after admission.
potassium dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, potassium dosage measured in mg/dl at admission and up to 48 hours after admission.
chlorine dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution,chlorine dosage measured in mg/dl at admission and up to 48 hours after admission.
alanine transferase dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, alanine transferase dosage measured in mg/dl at admission and up to 48 hours after admission.
lactic dehydrogenase dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, lactic dehydrogenase dosage measured in mg/dl at admission and up to 48 hours after admission.
sodium dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, sodium dosage measured in mg/dl at admission and up to 48 hours after admission.
creatinine dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, creatinine dosage measured in mg/dl at admission and up to 48 hours after admission.
c | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution, creatinine dosage measured in mm³ at admission and up to 48 hours after admission.
total and fractions bilirubin dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory tests and their evolution: urea, creatinine, uric acid, sodium, potassium and chlorine, lactic dehydrogenase (DHL), aspartate transferase (AST), alanine transferase (ALT), total and fractions bilirubin and platelets;
uric acid dosage | from admission in the hospital until 48 hours after delivery
  Baseline laboratory test and the evolution. urea, creatinine, uric acid, sodium, potassium and chlorine, lactic dehydrogenase (DHL), aspartate transferase (AST), alanine transferase (ALT), total and fractions bilirubin and platelets;
Evolution of blood pressure in the puerperium | from 24 after delivery to 48 hours
  Evolution of blood pressure in the puerperium
Number of hypertensive peaks | from 24 after delivery until discharge of the hospital
  Number of hypertensive peaks (systolic blood pressure of 180mmHg and/or diastolic blood pressure of 120mmHg);
need for maintenance antihypertensive treatment | from 24 after delivery until discharge of the hospital
  Identify the presence or absence of maintenance antihypertensive drugs
number of antihypertensive drugs; | from 24 after delivery until discharge of the hospital
  quantify how many antihypertensive medications are being used
Allergic reactions | from 24 after delivery to 48 hours
  Questionnaire with options for allergic manifestations: urticaria, angioedema, eczema, asthma.
Gastrointestinal side effects | from 24 after delivery to 48 hours
  Questionnaire with options for acute gastrointestinal effects: abdominal pain, dyspepsia and diarrhea
Time between postoperative and unassisted ambulation | from 24 after delivery to 48 hours
  Time between postoperative and unassisted ambulation
Length of hospital stay | From hospital admission to hospital discharge date or up to eight days after surgery whichever comes first.
  Length of hospital stay
Compound maternal morbidity | from 24 after delivery until discharge date or up to eight days after surgery whichever comes first.
  Compound maternal morbidity (eclampsia, acute pulmonary edema, HELLP syndrome, difficult-to-control hypertension, intracranial hemorrhage, renal failure and others);
Maternal death | from 24 after delivery until discharge date or up to eight days after surgery whichever comes first.
  Space reserved in the questionnaire to be described according to the death certificate the primary cause of maternal death.
Costs related to analgesic medications | from 24 after delivery until discharge date or up to eight days after surgery whichever comes first.
  Accounting for the cost related to each dose doses of anesthetic medications that were used in addition to the therapeutic regimens of the experiment were used

CONTACTS AND LOCATIONS:
Locations (1):
- IMIP, Recife, Pernambuco, Brazil